CLINICAL TRIAL: NCT00858273
Title: Regulation of Glutathione Homeostasis in Adolescents With Type 1 Diabetes - Study B
Brief Title: Glutathione Metabolism in Adolescents With Type 1 Diabetes - Study B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: JDRF 1-2006-627-B
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Glutathione
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antioxidant Supplement (Active Comparator): Vitamin C 250 mg; beta-carotene 6 mg; vitamin E 30 mg; selenium 100 mcg; zinc 20 mg
  Interventions: Dietary Supplement: Antioxidant supplement; Other: Diabetes treatment; Drug: Regular Insulin
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Antioxidant supplement; Other: Diabetes treatment; Drug: Regular Insulin

INTERVENTIONS:
Dietary Supplement: Antioxidant supplement — 1 capsule daily with dinner
Other: Diabetes treatment — Intensification of diabetes treatment regimen, including education and counseling, home blood glucose monitoring, multiple daily insulin injections (MDI), diet plan, and frequent phone contact with a certified diabetes educator
Drug: Regular Insulin — Regular Insulin, IV, to maintain blood glucose in normoglycemic range (70-140) during metabolic study

SUMMARY:
Glutathione is normally present at high levels in the blood and plays an important role in the body's defense against oxidative stress, that is, against the damage caused to the body by several reactive oxygen species produced by the metabolism of most nutrients, including glucose. Glutathione is a small peptide made from 3 amino acids, glutamate, cysteine, and glycine.

This study is looking at how blood sugar levels may affect the way glutathione is made and used by the body. Since glutathione is continuously synthesized and broken down, the amount of glutathione present in the blood depends on the balance between its rate of synthesis and its rate of use.

In earlier studies, we found that in poorly controlled diabetic teenagers, glutathione was low, not because it was not produced fast enough, but because it was used at an excessive rate. In this study, we want to find out whether improving blood sugar control will increase glutathione levels, and, if so, how long this will take. We also hope to find out if oral supplementation with a mixture of several antioxidant vitamins and minerals will increase glutathione levels more than taking a placebo.

DETAILED DESCRIPTION:
Forty adolescents with T1D will undergo a measurement of blood glutathione concentration and markers of oxidative stress (plasma protein-bound 3-nitrotyrosine, and urinary 8OH-2-dG, and F2-isoprostane excretion, markers of oxidative damage to protein, DNA and lipids, respectively) while at near normoglycemia, on two separate occasions:

* first, when in poor glucose control (HbA1c>7.5%); and
* secondly, after 3 to 9 months months of improved blood glucose control, along with the administration of either a placebo, or a mixture of antioxidant minerals and vitamins based on a randomization scheme.

Between the two metabolic study days, patients will receive the same intensified diabetes regimen consisting of education and counseling, home blood glucose monitoring, multiple daily insulin injections (MDI), diet plan, and frequent phone contact with a certified diabetes educator.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes, using usual criteria such as: glycosuria, hyperglycemia prior to treatment
* BMI <25 kg/m2
* Age 12-21
* HbA1c>7.5%
* No evidence of diabetic complications
* Written informed consent from parents or legal guardian, and assent from patient

Exclusion Criteria:

* Presence of significant anemia (hemoglobin <11g/dL)
* Presence of intercurrent illness such as infection
* Presence of chronic disease such as other endocrine deficiency, chronic respiratory or cardiac disease
* Chronic use of medication other than insulin
* Use of vitamin or mineral supplements within 2 weeks of study

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Darmaun, MD, PhD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Benson M, Hossain J, Darmaun D. Improved glycemic control either alone, or combined with antioxidant supplementation, fails to restore blood glutathione or markers of oxidative stress in adolescents with poorly controlled type 1 diabetes. Nutr Res. 2023 Sep;117:83-90. doi: 10.1016/j.nutres.2023.05.010. Epub 2023 May 25. PMID 37515943

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antioxidant Supplement | Placebo
Started | 20 | 20
Completed | 17 | 15
Not Completed | 3 | 5
Not completed — Protocol Violation | 3 | 5

BASELINE CHARACTERISTICS:
Population: 8 of the 40 Participants were not eligible for the second admission to the CRC due to the inability to drop their HbA1C by 0.5% within the time frame of the project. Therefore, 32 Participants were used for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Antioxidant Supplement | Placebo | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 15 | 32
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (2.3) | 15.8 (2.6) | 15.8 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 14 | 12 | 26
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Glutathione Concentration
Description: While at near normoglycemia
Time Frame: After 3-9 months of improved blood glucose control (HbA1c decrease of >0.5%)
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Antioxidant Supplement | Placebo
Number analyzed (Participants) | 17 | 15
umol/L | 706 (236) | 734 (215)

2. Secondary Outcome: Plasma Protein Bound 3-nitrotyrosine
Description: Marker of oxidative stress
Time Frame: After 3-9 months of improved blood glucose control (HbA1c decrease of >0.5%)
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Antioxidant Supplement | Placebo
Number analyzed (Participants) | 17 | 15
ng/mL | 4.26 [1.65 to 19] | 7.13 [1.22 to 10.9]

ADVERSE EVENTS:
Arm/Group | Antioxidant Supplement | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/17 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes